CLINICAL TRIAL: NCT02682862
Title: Effects of Ultra-long Acting Bronchodilator Therapy Assessed by Impulse Oscillometry in Smoking Asthmatics Taking Inhaled Corticosteroids
Brief Title: Ultra-long Acting Bronchodilator Therapy in Smoking Asthmatics
Acronym: MAN05
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2013RC06; 2014-005317-23 (EudraCT Number)
Record Dates: First submitted 2016-02-04; First posted 2016-02-17 (Estimated); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Asthma
Keywords: tiotropium; olodaterol; smoker; cigarette; bronchodilator
MeSH Terms: conditions — Asthma | interventions — Tiotropium Bromide; tiotropium-olodaterol; olodaterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spiolto Respimat (Experimental): olodaterol hydrochloride 2.5mcg, tiotropium bromide 2.5mcg 2 puffs OD (once daily) for 2-4 weeks. Participants then enter washout period and receive alternative treatment arm
  Interventions: Drug: olodaterol hydrochloride 2.5mcg, tiotropium bromide 2.5mcg
- Striverdi Respimat (Active Comparator): olodaterol 2.5mcg 2 puffs OD (once daily) for 2-4 weeks. Participants then enter washout period and receive alternative treatment arm
  Interventions: Drug: olodaterol 2.5 mcg

INTERVENTIONS:
Drug: olodaterol hydrochloride 2.5mcg, tiotropium bromide 2.5mcg — Inhaler: 2.5 microgram tiotropium (as bromide monohydrate) and 2.5 microgram olodaterol (as hydrochloride) per puff. 2 puffs once daily
  Other Names: Spiolto Respimat 2.5mcg/2.5mcg
  Arms: Spiolto Respimat
Drug: olodaterol 2.5 mcg — Inhaler: 2.5 microgram Olodaterol (as hydrochloride) per puff. 2 puffs once daily
  Other Names: Striverdi Respimat 2.5mcg
  Arms: Striverdi Respimat

SUMMARY:
Single centre, open-label, random order, cross-over trial, recruited over a period of approximately 2 years. Sufficient participants enrolled to complete 16 adults. Withdrawn subjects may be replaced.

This clinical trial will assess the effects of ultra-long acting bronchodilator therapy in smoking asthmatics taking inhaled corticosteroids. This will be via a pulmonary function test called impulse oscillometry.

DETAILED DESCRIPTION:
Cigarette smoking in asthma is associated with poorer asthma control and a higher frequency of asthma attacks. Despite this, smoking cessation rates are very low due to the highly addictive nature of tobacco smoking. Asthma in smokers is particularly challenging to manage because it is resistant to the beneficial effects of inhaled corticosteroids, the main treatment for asthma.

Unfortunately, there is no guideline consensus regarding how to best manage asthmatics who smoke. Research studies in asthma tend to exclude smokers because of concerns about recruiting patients with chronic obstructive pulmonary disease (COPD). Hence, there is an unmet need for research studies in asthmatics who are unable to stop smoking.

In view of the above, we propose to assess the effects of two different types of bronchodilators (inhalers which help open up the airways), in asthmatics who continue to smoke.

Participants will receive both of the following drugs for 2-4 weeks in random order, with a 2-3 week washout period in between:

Olodaterol which is a new long-acting bronchodilator. Olodaterol combined with tiotropium (dual bronchodilators). We wish to compare these inhalers using a sensitive pulmonary function test called impulse oscillometry.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers aged 18-65 years with persistent asthma and on inhaled corticosteroids (at least 400 micrograms beclomethasone dipropionate equivalent dose daily)
* Current smoker
* Forced Expiratory Volume in 1 second (FEV1) ≥ 60 % predicted
* Ability to give informed consent
* Agreement for their General Practitioner to be made aware of study participation and to receive feedback as relevant to the participant's well being

Exclusion Criteria:

* Other significant respiratory diseases, in the opinion of the investigator, such as COPD or bronchiectasis.
* An asthma exacerbation or respiratory tract infection requiring systemic steroids and/or antibiotics within 1 month of the study commencement or 3 months if hospital admission was required
* Any clinically significant medical condition that may endanger the health or safety of the participant
* Participation in another drug trial within 30 days before the commencement of the study
* Pregnancy or lactation
* Unable to comply with the procedures of the protocol
* Unable or unwilling to consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2019-05-22 (Actual)

PRIMARY OUTCOMES:
Airway resistance at 5Hz (R5) | 2-4 weeks
  measured by Impulse oscillometry (IOS)

SECONDARY OUTCOMES:
RF | 2-4 weeks
  Impulse Oscillometry: Resonant Frequency
X5 | 2-4 weeks
  Impulse Oscillometry: Reactance at 5Hz
AX | 2-4 weeks
  Impulse Oscillometry: Reactance Area
R5-R20 | 2-4 weeks
  Impulse Oscillometry: Resistance at 5Hz minus Resistance at 20Hz, equating to small airway resistance
R20 | 2-4 weeks
  Impulse Oscillometry: Resistance at 20Hz
FEF25-75 pre and post challenge | 2-4 weeks
  Spirometry: Forced expiratory flow 25%-75% pre and post bronchial challenge (assessing change)
FVC pre and post challenge | 2-4 weeks
  Spirometry: Forced vital capacity pre and post bronchial challenge (assessing change)
FEV1 pre and post challenge | 2-4 weeks
  Spirometry: Forced expiratory volume in 1 second pre and post bronchial challenge (assessing change)
Mannitol PD30 | 2-4 weeks
  Provocation dose of mannitol causing 30% increase in R5
Mannitol RDR | 2-4 weeks
  Response-Dose Ratio
R5 at PD30 | 2-4 weeks
  Airway Resistance at 5 Hertz at PD30
Salbutamol recovery time following mannitol challenge | 2-4 weeks
Domiciliary PEF | 2-4 weeks
  Peak Expiratory Flow
ACQ | 2-4 weeks
  Asthma Control Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sunny Jabbal, Mb Chb, Principal Investigator — University of Dundee; Brian Lipworth, MD, Mb Chb, Principal Investigator — University of Dundee
Locations (1):
- Scottish Centre for Respiratory Research, University of Dundee, Ninewells Hospital and Medical School, Dundee, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lipworth B, RuiWen Kuo C, Jabbal S, Chan R. Inhaled triple therapy and airway hyperresponsiveness in persistent asthma. Ann Allergy Asthma Immunol. 2021 May;126(5):597-598. doi: 10.1016/j.anai.2021.01.032. Epub 2021 Feb 3. No abstract available. PMID 33548471
- [Derived] Jabbal S, Kuo CR, Lipworth B. Randomized controlled trial of triple versus dual inhaler therapy on small airways in smoking asthmatics. Clin Exp Allergy. 2020 Oct;50(10):1140-1147. doi: 10.1111/cea.13702. Epub 2020 Jul 27. PMID 33180376